CLINICAL TRIAL: NCT07391800
Title: Single-Arm Study of Compound Granules of Hedyotis Diffusa for Chronic Atrophic Gastritis
Brief Title: Compound Granules of Hedyotis Diffusa for Chronic Atrophic Gastritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Liao Yun, Chief Pharmacist, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYun
Record Dates: First submitted 2025-12-23; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Chronic Atrophic Gastritis With Hyperplasia (Diagnosis)
Keywords: Compound Granules of Hedyotis diffusa; chronic atrophic gastritis
MeSH Terms: conditions — Disease; Gastritis, Atrophic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compound Granules of Hedyotis diffusa Group (Experimental): Patients received Compound Granules of Hedyotis diffusa for 12 months, followed by a 12-month follow-up period.
  Interventions: Drug: Compound Granules of Hedyotis diffusa

INTERVENTIONS:
Drug: Compound Granules of Hedyotis diffusa — 12-month treatment with Compound Granules of Hedyotis diffusa and 12-month follow-up

SUMMARY:
Chronic atrophic gastritis is considered a premalignant lesion of gastric cancer. The development of gastric cancer usually follows the Correa sequence: chronic superficial gastritis → chronic atrophic gastritis → intestinal metaplasia → dysplasia → gastric cancer. Premalignant lesions of gastric cancer, such as superficial gastritis with intestinal metaplasia, atrophic gastritis with intestinal metaplasia, and atypical hyperplasia, have a high risk of progressing to gastric cancer if not intervened in a timely and effective manner. Currently, Western medicine treatment for chronic atrophic gastritis mainly includes eradicating Helicobacter pylori, supplementing folic acid or vitamins, and using gastric mucosal protectants. However, there is no specific drug to reverse gastric mucosal atrophy, and clinical needs are far from being met.

According to traditional Chinese medicine (TCM) theory, chronic atrophic gastritis falls into the categories of "epigastric pain" and "gastric discomfort". It is treated based on syndrome differentiation, including various syndrome types such as spleen-stomach deficiency, qi stagnation and blood stasis, and damp-heat accumulation. TCM compound preparations have shown unique advantages in the treatment of chronic atrophic gastritis due to their advantages of multi-target and overall regulation. Chinese patent medicines such as Moluo Dan and Weifuchun Capsules have effects such as clearing heat and detoxifying, anti-inflammation, anti-bacteria, and treating chronic gastritis. Their clinical application provides important references for TCM intervention in chronic atrophic gastritis. However, there are still problems such as large individual differences in efficacy and poor response in some patients. Moreover, the precise treatment strategies for different TCM syndrome types (such as spleen-stomach deficiency type and liver-stomach disharmony type) need to be optimized.

Compound Granules of Hedyotis diffusa, composed of three TCM herbs: Hedyotis diffusa, Smilax china L., and Solanum lyratum Thunb., is a classic ancient prescription that has been used in Shanghai First People's Hospital for many years. It is a hospital preparation approved for production by the Shanghai Food and Drug Administration (Approval No.: SYZ-ZF-003-2007), with the effects of clearing heat and detoxifying, and resolving blood stasis and dissipating masses. It is used for superficial gastritis, atrophic gastritis with intestinal metaplasia, atypical hyperplasia, etc., and has a preventive and therapeutic effect on premalignant lesions of gastric cancer and gastric cancer. Long-term clinical observations have found that it can not only relieve symptoms but also may have a certain improvement effect on the pathological changes of gastric mucosa.

Literature reports indicate that traditional Chinese medicines represented by Hedyotis diffusa, Smilax china L., and Solanum lyratum Thunb. have good anti-inflammatory and anti-tumor activities. Due to differences between Chinese and Western cultures and the complex composition of TCM, TCM and TCM compound preparations have not yet been universally recognized by the international community. Therefore, studying TCM compound preparations using modern scientific methods, clarifying their effects as much as possible, and endowing traditional medicine with modern scientific connotations hold great clinical and social significance.

Long-term clinical practice observations in Shanghai First People's Hospital have found that Compound Granules of Hedyotis diffusa has a certain preventive and therapeutic effect on atrophic gastritis with intestinal metaplasia and premalignant lesions of gastric cancer. However, there is currently a lack of systematic clinical research data support. Therefore, this clinical study will comprehensively evaluate the efficacy and safety of Compound Granules of Hedyotis diffusa in the treatment of atrophic gastritis, so as to provide a basis for its clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 and 80 years old;
* Diagnosed with atrophic gastritis with intestinal metaplasia by gastroscopic examination and histopathological diagnosis;
* TCM diagnosis of spleen-stomach damp-heat syndrome;
* Able to understand and sign the informed consent form, and willing to cooperate to complete the entire research process.

Exclusion Criteria:

* Previous history of gastric cancer or complicated with high-grade intraepithelial neoplasia;
* Lactation or pregnancy;
* Severe mental illness;
* Other severe systemic diseases (such as malignant tumors, severe heart, liver, or renal failure, etc.).

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic Diagnosis | One year after enrollment
  Improvements in histologic scores and effective rates were calculated in patients who had undergone biopsy at least 2 times at the same site before and after treatment. Improved efficacy of histology was rated as effective or ineffective. Effective was defined as atrophy or intestinal metaplasia (IM) decreased at least one grade. Ineffective was defined as no improvement or the condition becoming worse.

SECONDARY OUTCOMES:
Endoscopic Assessment | One year after enrollment
  A senior endoscopist blinded to the patients' treatment group assignment scored the endoscopic findings in accordance with the Kyoto Classification of Gastritis (Appendix 3, Supplemental Digital Content 1, http://links.lww.com/JCG/A802).

OTHER OUTCOMES:
Symptom | A follow-up visit was conducted at baseline and at 4, 13, 26, 39, and 52 weeks following drug administration.
  Symptom improvement efficacy was categorized into three grades: markedly effective (complete or near-complete resolution of clinical symptoms including epigastric pain, abdominal distension, anorexia, belching, and acid regurgitation); effective (significant symptom relief or >50% reduction in symptom scores); and ineffective (<50% reduction in symptom scores or symptom exacerbation). Total effective rate was calculated as the percentage of the sum of markedly effective and effective cases relative to the total cases.
Adverse Event Incidence Rate | A follow-up visit was conducted at 4, 13, 26, 39, and 52 weeks following drug administration.
  An independent investigator interviewed patients quarterly to record adherence and queried about adverse events.
Serum Gastric Function Parameters | A follow-up visit was conducted at baseline and at 4, 13, 26, 39, and 52 weeks following drug administration.
  Serum gastric function indicators were tested every three months via blood sampling, with the detection of Pepsinogen 1 (PGⅠ) and Pepsinogen 2 (PGⅡ).

CONTACTS AND LOCATIONS:
Overall Officials: Yun Liao, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No